CLINICAL TRIAL: NCT06151678
Title: An Evaluation of a Public Health Campaign Related to Persistent Pain in the United Kingdom
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Collaborators: Prof Denis Martin (Unknown); Prof Cormac Ryan (Unknown); Gail Sowden (Unknown); Prof Lorimer Moseley (Unknown); Dr Jonathan Emerson (Unknown)
Responsible Party: Principal Investigator, Nick Livadas, Senior Lecturer, Teesside University
Other Study IDs: TeessideUniversitySOHLS
Record Dates: First submitted 2022-12-18; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Pain, Chronic; Pain, Back; Musculoskeletal Pain; Arthritis; Back Pain
Keywords: Persistent Pain; Public Health
MeSH Terms: conditions — Chronic Pain; Back Pain; Musculoskeletal Pain; Arthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- UK population survey: The UK population who accessed the electronic survey link disseminated via social media and via a gatekeeper at a Scottish council
- Participants attending online webinars: Individuals who signed up for an online webinar related to persistent pain. This group offered quantitative feedback via online surveys and qualitative data via interview.
  Interventions: Other: Pain Education
- Participants who attended in person seminars during a community outreach tour: Individuals who attended six different venues across the English county of Lincolnshire. This group offered quantitative feedback via paper and online surveys and qualitative data via interview.
  Interventions: Other: Pain Education
- Brain bus cohort: Participants who attended a pop up interactive tent with practical demonstrations to improve pain related knowledge. This group offered quantitative feedback via paper postcards and qualitative data via interview.
  Interventions: Other: Pain Education
- Community outreach tour volunteers: Focus groups were arranged for those who volunteered to lead and deliver the community outreach tour

INTERVENTIONS:
Other: Pain Education — Pain education was offered to health professionals and the general public using with a focus on pain neuroscience. This was offered with a lecture from pain scientists, personal reflections from individuals with lived experience and health care professionals.
  Groups: Brain bus cohort; Participants attending online webinars; Participants who attended in person seminars during a community outreach tour

SUMMARY:
The goals of this study are

* To define what the public perceptions of persistent pain using a national survey
* Explore relationships between the reported pubic beliefs and demographic factors collected.
* To evaluate the impact of a public health campaign to increase awareness of persistent pain and develop understanding of pain that aligns with contemporary science.

DETAILED DESCRIPTION:
This study included a cross sectional survey of the UK population to understand what the beliefs are regarding persistent pain. This survey will be distributed electronically using social media and to a Scottish council. Differences in beliefs will be explored using the demographic data collected.

The second aspect of the study is the evaluation of a public health campaign called 'Flippin Pain'. This study component included the evaluation of online webinars with pre, post, 3 month, 6 month and 12 month longitudinal data collection. One of the online seminars also included the qualitative evaluation using semi structured interviews.

The third part of the study was the evaluation of a community outreach tour in the county of Lincolnshire, United Kingdom. This included the collection of pain belief data before an in person seminar, immediately afterwards, then at 3 months. Semi structured interviews were also conducted with participants who attended the webinars. As part of the outreach tour an interactive pop up tent gave members of the public an understanding of pain using practical demonstrations. The was evaluated using short semi structured interviews along with written summaries offered by the participants before and immediately after experiencing the practical demonstrations.

After the community outreach tour, two focus groups were conducted with the campaign volunteers with an aim to understand the experience of those involved. The focus groups asked the participants to reflect on the successes and challenges of delivering a community based public health outreach tour.

ELIGIBILITY:
Inclusion Criteria:

* UK cross sectional survey - All adults over the age of 18 who are the capable of offering informed consent)
* Online webinar study - Adults over the age of 18 who attend an online webinar related to persistent pain
* Community outreach tour seminar - Adults over the age of 18 who attend an in person seminar
* Brain Bus - Adults over the age of 18 who experience the interactive demonstrations relating to persistent pain
* Focus Groups - Volunteers who participated in the Flippin Pain community outreach tour within the county of Lincolnshire

Exclusion Criteria:

* Individuals younger than 18 years of age.
* For the cross sectional UK survey, adults who lived outside of the UK were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cross sectional survey - Adults over the age of 18 that respond to an electronic survey link posted on FaceBook groups and employees of a Scottish council.
  Webinars and Seminars - Individuals who attended an education webinar or seminar related to persistent pain.
  Brain Bus - Individuals who engaged in the interactive experience to learn about persistent pain.
  Focus Groups - A total of 20 volunteers who supported the community outreach tour in the English county of Lincolnshire.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Pain Beliefs Questionnaire | Used within the cross sectional survey and pre and post webinars and seminars. This has been administered immediately before the webinar or seminar, immediately after the webinar or seminar, then at 3 month, 6 month and 1 year.
  A validated survey to ascertain pain beliefs from the general population

SECONDARY OUTCOMES:
HC-PAIRS | This is administered online immediately prior to adttendance of an online webinar. Immediately after the webinar. Then further administration at 3 month, 6 month and 1 year.
  A validated survey to ascertain the pain beliefs of healthcare professionals.
Osteoarthritis Conceptual Scale | This is administered online immediately prior to attendance of an online webinar. Immediately after the webinar. Then further administration at 3 month, 6 month and 1 year.
  A 33 item survey to ascertain beliefs regarding knee osteoarthritis

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data may be shared from the survey responses.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When the evaluation is completed and submitted to a peer review journal. Estimated 2024.
Access Criteria: Additional data beyond what is included in the results section of the manuscript can be made available within the supplementary files.